CLINICAL TRIAL: NCT04653857
Title: Evaluation of Cardiological Tests Before Returning to Sport in Athletes After COVID-19 Infection (CADE Study)
Brief Title: Cardiac Assessment After Covid-19 Disease in Elite Altheltic Population
Acronym: CADE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Clinique du Millenaire (Other); Centre Hospitalier Universitaire de Nīmes (Other); Centre hospitalier de Perpignan (Other); ligue nationale de Basket (Unknown); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0648
Record Dates: First submitted 2020-12-03; First posted 2020-12-04 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: High-level athlete; recent COVID 19 infection, symptomatic or not
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-level athlete who had a recent COVID 19 infection, symptomatic or not: High-level athlete who had a recent COVID 19 infection, symptomatic or not

SUMMARY:
COVID-19 infection coud induce cardiac injuries. Before returning to sport, cardiac evaluation is recommended by sports federations, based on the precautionary principle and the opinion of expert consensus.

The aim of this study is to to determine the prevalence of abnormalities in cardiological examinations realized in athletes who have suffered from COVID-19 infection, symptomatic or not.

DETAILED DESCRIPTION:
Cardiac injuries linked to COVID-19 infection are frequently described in symptomatic and hospitalized people and are associated with a poorer prognosis. The question of possible myocardial damage in people without or moderately symptomatic is less established. The presence of a myocarditis associated with COVID-19 infection is a key issue for the sports cardiologist since this cardiac inflammation may be associated with an increased risk of sudden death in the athlete.

In absence of scientific data and on the basis of the precautionary principle, the ministry (Guide to health recommendations for sports resumption, Sports French Ministry, May 2020), sports federations and certain expert consensus have proposed in May 2020 after being released from lockdown, algorithms for carrying out systematic cardiac examinations before resuming intense sport (professional or high-level athletes). These algorithms typically provide a comprehensive cardiac assessment with resting ECG, resting echocardiography, and maximal exercice test. The performance of cardiac MRI, the most sensitive exam for detecting possible myocarditis, remains at the discretion of the cardiologist depending on the interpretation of the first examinations.

Given a much larger screening for COVID-19 infection than in March, with the performance of virological PCR tests required weekly by certain sports federations, the prevalence of COVID-19 infection is important in the athletic population, mostly in a- or pauci-symptomatic athletes. In case of positivity, a cardiac evaluation is therefore often recommended.

The aim of this study is to determine the prevalence of cardiac abnormality encountered during cardiac examinations performed in athletes before resuming intense sport, after infection with COVID-19.

The target population is High-level athlete (professionals or high-level ministerial list), who had a recent COVID 19 infection, symptomatic or not

To perform this study, the investigators will use existing data from patients' medical records (March 2019, March 2021). Anonymized data will be provided to the methodological team for analysis. The data will be kept for 2 years after publication. The data collected will be :

* the sport practiced
* Age and sex
* Date of positive PCR
* Classification of the symptom intensities related to COVID-19 infection: (asymptomatic, mild symptoms, moderate symptoms, cardiac symptoms)
* 12-lead resting electrocardiogram (heart rate, interpretation by the cardiologist, anomaly or not)
* Maxmal exercice test (maximum heart rate, maximum power or speed, oxygen saturation, presence of arrhythmia or not)
* Resting echocardiography (LVEF, overall LV longitudinal strain, abnormal or not in segmental kinetics, presence or not of pericardial effusion)
* MRI (if done): LVEF, presence of an abnormality or not, in particular late enhancement
* Holter ECG if done (presence or not of arrhythmia)
* Biology if done (increase or not in troponin or D-Dimers

ELIGIBILITY:
Inclusion criteria:

* High-level athlete
* recent COVID 19 infection, symptomatic or not
* evidence of COVID 19 infection by PCR or serology

Exclusion criteria:

- subject opposition

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High-level athlete (professionals or high-level ministerial list) who had a recent COVID 19 infection, symptomatic or not
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiac abnormality | 1 to 3 weeks after COVID-19 infection
  Prevalence of cardiac abnormality encountered during examinations performed in athletes before resuming intense sport, after infection with COVID-19

SECONDARY OUTCOMES:
Demographic variables | 1 to 3 weeks after COVID-19 infection
  Demographic variables associated with detected cardiac abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane CADE, MD, Principal Investigator — Clinique du Millenaire, Montpellier, France; Christophe HEDON, MD, Study Director — UH MONTPELLIER
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC